CLINICAL TRIAL: NCT05448378
Title: Evaluation of the Effects of D-chiro-inositol in Female Healthy Volunteer
Brief Title: Evaluation of D-chiro-inositol Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lo.Li.Pharma s.r.l (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DCI-Evaluation
Record Dates: First submitted 2022-07-04; First posted 2022-07-07 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-07

CONDITIONS: Inositol; Testosterone; Insulin; Ovulation; Asprosin
MeSH Terms: conditions — Insulin Resistance; Arachnodactyly

STUDY DESIGN:
Intervention Model Description: Human healthy women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-chiro-inositol (Experimental): Patients will take D-chiro-inositol. We will make two blood sampling, at the baseline and after one-month treatment
  Interventions: Dietary Supplement: D-chiro-inositol

INTERVENTIONS:
Dietary Supplement: D-chiro-inositol — D-chiro-inositol 600 mg twice per day on an empty stomach for one month

SUMMARY:
Healthy women will take tablets containing 600 mg D-chiro-inositol twice per day for one month. We will evaluate metabolic and hormonal.parameters, as insulienmia, glycemia, estradiol, testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Good state of health;
* Regular menstrual cycle.

Exclusion Criteria:

* pregnancy;
* delivery in the previous 6 months;
* currently breastfeeding;
* menopause;
* alcohol or drug abuse;
* insulin resistance defined as HOMA-IR index greater than or equal to 2.5;
* other medical morbidities, such as hypertension, PCOS, or diabetes;
* oligomenorrhea or amenorrhea;
* current treatment with corticosteroids or hormones (oral contraceptives, estrogensic, progestogensin);
* use of GnRH analogues, SERMs, or SPRMs within the previous 6 months.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
Testosterone | 30 days
  Serum values of testosterone

SECONDARY OUTCOMES:
BMI | 30 days
  body-mass index
Glycemia | 30 days
  Serum values of glucose
Insulinemia | 30 days
  Serum values of insulin
HOMA-IR index | 30 days
  Model of assessment for insulin resistance
FSH | 30 days
  Serum values of FSH
LH | 30 days
  Serum values of LH
Estradiol | 30 days
  Serum values of estradiol
DHEAS | 30 days
  Serum values of DHEAS
Asprosin | 30 days
  Serum values of asprosin

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - ASL Civitavecchia, Rome, Lazio
  - ALMA RES, Rome, Lazio

IPD SHARING:
Plan to Share IPD: No